CLINICAL TRIAL: NCT03421743
Title: An Open-label, Non-controlled, Multicentre, Pilot Clinical Trial of Inhaled Molgramostim in Subjects With Antibiotic-resistant Non-tuberculosis Mycobacterial (NTM) Infection
Brief Title: Pilot Trial of Inhaled Molgramostim in Non-tuberculous Mycobacterial (NTM) Infection
Acronym: OPTIMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Savara Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAV008-01; 2017-003374-14 (EudraCT Number)
Record Dates: First submitted 2018-01-16; First posted 2018-02-05 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2023-03

CONDITIONS: Mycobacterium Infections, Nontuberculous
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous

STUDY DESIGN:
Intervention Model Description: Open-label, non-controlled, multicenter, pilot clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhaled molgramostim/antimycobacterials (Experimental): Inhaled molgramostim administered in participants who remain sputum culture positive while currently on a multidrug NTM guideline-based antimycobacterial regimen, which has been ongoing for at least 6 months prior to the Baseline Visit
  Interventions: Drug: Inhaled molgramostim; Drug: Antimycobacterial regimen
- Inhaled molgramostim (Experimental): Inhaled molgramostim administered in participants who remain sputum culture positive but have stopped a multidrug NTM guideline-based antimycobacterial regimen at least 28 days prior to Screening due to lack of response or intolerance, or who never started such treatment
  Interventions: Drug: Inhaled molgramostim

INTERVENTIONS:
Drug: Inhaled molgramostim — 300 µg / dose molgramostim (recombinant human GM-CSF) for inhalation
  Other Names: rh-GM-CSF
Drug: Antimycobacterial regimen — Multidrug NTM guideline-based antimycobacterial regimen
  Arms: Inhaled molgramostim/antimycobacterials

SUMMARY:
The trial is an open-label, non-controlled, multicenter, pilot clinical trial of inhaled molgramostim (recombinant human granulocyte-macrophage colony stimulating factor; rhGM-CSF) in subjects with persistent pulmonary non-tuberculous mycobacterial (NTM) infection. Participants will be treated for 24-weeks with inhaled molgramostim and followed up for 12-weeks after end of treatment. The primary aim of the trial is to investigate the efficacy of inhaled molgramostim on NTM sputum culture conversion to negative.

DETAILED DESCRIPTION:
The study will comprise a Screening Visit, a Baseline Visit, a 24-week treatment period and a 12-week follow-up period. 30 adult participants with a history of chronic NTM infection with at least 2 positive cultures in the prior 2 years, of which at least one is within the last 6 months prior to Screening, will be considered for enrollment. Participants should provide a positive NTM sputum culture at Screening to be eligible.

Two subgroups of participants will be recruited:

* Group 1: Participants who remain sputum culture positive while currently on a multidrug NTM guideline based antimycobacterial regimen, which has been ongoing for at least 6 months prior to the Baseline Visit.
* Group 2: Participants who remain sputum culture positive but have either stopped a multidrug NTM guideline based antimycobacterial regimen at least 28 days prior to Screening due to lack of response or intolerance, or never started such treatment.

The treatment period will consist of 14 trial visits (Screening [within 10 weeks of Baseline], Baseline, and every 4 weeks to Week 48 [visits at Weeks 28, 36 and 44 included telephone contact, others included clinic visits]) and a Follow-up visit 12 weeks after the end of treatment.

At the Baseline visit, eligible participants will start treatment with molgramostim nebulizer solution, 300 μg, administered by inhalation using an eFlow Nebulizer System. At each visit, sputum samples will be collected for staining and microscopy, and microbiological culture. In addition, clinical assessments including body weight, patient reported outcomes, and diffusion capacity of the lung for carbon monoxide (DLCO) will be conducted at each clinic visit. Spirometry will be assessed at Baseline, and at Weeks 12, 24, 32, 40 and 48. A 6-minute walk test (6-MWT) will be conducted at Baseline, at Weeks 12, 24, 48 and at the 12-week Follow-up visit. Safety laboratory samples will be collected at Screening, Baseline and at Weeks 4, 12, 24, 32, 40, 48 and at the 12-week Follow-up visit. Anti-GM-CSF antibodies will be assessed at Baseline, at Week 4, 12, 24, 32, 48, and at the 12-week Follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. History of chronic pulmonary infection with MAC or M. abscessus (defined as at least 2 documented positive sputum cultures in the prior 2 years, of which at least one was obtained in the 6 months prior to Screening).
2. Subject fulfills one of the following criteria:

   * Subjects who remain sputum culture positive while currently on a multidrug NTM guideline based antimycobacterial regimen, which has been ongoing for at least 6 months prior to the Baseline Visit
   * Subjects who remain sputum culture positive but have either stopped a multidrug NTM guideline based antimycobacterial regimen at least 28 days prior to Screening due to lack of response or intolerance, or never started such treatment.
3. Ability to produce at least 2 mL of sputum or be willing to undergo an induction that produces at least 2 mL of sputum for clinical evaluation.
4. Female or male ≥18 years of age.
5. Females who have been post-menopausal for more than 1 year or females of childbearing potential after a confirmed menstrual period using a highly efficient method of contraception (i.e. a method with less than 1% failure rate such as combined hormonal contraception, progesterone-only hormonal contraception, intrauterine device, intrauterine hormone- releasing system, bilateral tubal occlusion, vasectomized partner, sexual abstinence), during and until thirty (30) days after last dose of trial treatment. Females of childbearing potential must have a negative serum pregnancy test at Screening (Visit 1) and a negative urine pregnancy test at dosing at Baseline (Visit 2) and must not be lactating.
6. Males agreeing to use condoms during and until thirty (30) days after last dose of medication, or males having a female partner who is using adequate contraception as described above.
7. Willing and able to provide signed informed consent.
8. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures specified in the protocol as judged by the investigator

Exclusion Criteria:

1. Subjects diagnosed with cystic fibrosis.
2. Prior therapy with inhaled or systemic GM-CSF.
3. Subjects with hemoptysis of ≥60 mL in a 24 hour period within 4 weeks prior to Screening.
4. Concurrent disease with a life expectancy of less than 6 months.
5. History of, or present, myeloproliferative disease, leukemia or other hematological malignancy.
6. Active pulmonary malignancy (primary or metastatic); or any malignancy requiring chemotherapy or radiation therapy within one year prior to Screening or anticipated during the study period.
7. Active allergic bronchopulmonary mycosis or connective tissue disease, inflammatory bowel disease or other autoimmune disorder requiring therapy associated with significant immunosuppression, such as systemic corticosteroids at a dose equivalent of 10 mg/day or more of prednisolone, within 3 months prior to Screening or anticipated during the study period.
8. Pulmonary tuberculosis requiring treatment or treated within 2 years prior to Screening.
9. HIV infection or other disease associated with significant immunodeficiency.
10. History of lung transplantation.
11. Any change in chronic NTM multi-drug antimycobacterial regimen within 28 days prior to Screening.
12. Treatment with any investigational medicinal product within 3 months of Screening.
13. Previous experience of severe and unexplained side-effects during aerosol delivery of any kind of medicinal product
14. Any other serious medical condition which in the opinion of the investigator would make the subject unsuitable for the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2020-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant Waterer, Prof., Principal Investigator — Royal Perth Hospital
Locations (5):
- Australia (4):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - The Prince Charles Hospital, Chermside West, Queensland
  - Greenslopes Private Hospital, Greenslopes, Queensland
  - Royal Perth Hospital, Perth, Western Australia
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomson RM, Loebinger MR, Burke AJ, Morgan LC, Waterer GW, Ganslandt C. OPTIMA: An Open-Label, Noncomparative Pilot Trial of Inhaled Molgramostim in Pulmonary Nontuberculous Mycobacterial Infection. Ann Am Thorac Soc. 2024 Apr;21(4):568-576. doi: 10.1513/AnnalsATS.202306-532OC. PMID 37948736

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study conducted in a total of 5 sites in Australia and the UK. First participant was enrolled on 1 March 2018 and last participant completed the study on 13 January 2020.
Pre-assignment Details: Adults with chronic pulmonary NTM infection and a positive sputum culture at Screening were recruited into 2 groups:
  1. On multidrug NTM guideline-based antimycobacterial regimen ongoing for ≥6 months prior to Baseline.
  2. Had stopped multidrug NTM regimen ≥28 days prior to Screening (lack of response/intolerance)/never started such treatment.
Groups:
- Inhaled Molgramostim/Antimycobacterials: Inhaled molgramostim administered in participants who remain sputum culture positive while currently on a multidrug NTM-guideline based antimycobacterial regimen, which has been ongoing for at least 6 months prior to the Baseline Visit
  Inhaled molgramostim: 300 µg / dose molgramostim (recombinant human GM-CSF) for inhalation
- Inhaled Molgramostim: Inhaled molgramostim administered in participants who remain sputum culture positive but have stopped a multidrug NTM-guideline based antimycobacterial regimen at least 28 days prior to Screening due to lack of response or intolerance, or who never started such treatment
  Inhaled molgramostim: 300 µg / dose molgramostim (recombinant human GM-CSF) for inhalation
Period: Overall Study
Arm/Group | Inhaled Molgramostim/Antimycobacterials | Inhaled Molgramostim
Started | 14 | 18
Completed | 11 | 16
Not Completed | 3 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: No "analysis sets" were defined. All participants were included in the analyses/data presentations, equivalent to a Full Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Molgramostim/Antimycobacterials | Inhaled Molgramostim | Total
Number analyzed (Participants) | 14 | 18 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 12 | 16
  >=65 years | 10 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (9.9) | 66.0 (9.0) | 66.6 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 2 | 8 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 16 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 2 | 0 | 2
  Australia | 12 | 18 | 30
NTM type [Count of Participants; unit: Participants] — Participants may have met one or more criteria
  Participants
    Mycobacterium avium complex | 11 | 13 | 24
    Mycobacterium abscessus | 3 | 6 | 9
Age at NTM diagnosis [Mean (Standard Deviation); unit: years] | 60.9 (9.7) | 60.1 (11.7) | 60.4 (10.7)
Smoking status [Count of Participants; unit: Participants]
  Never | 11 | 9 | 20
  Previous | 3 | 8 | 11
  Current | 0 | 1 | 1
Baseline Lower Respiratory Tract Infections - Visual Analogue Scale (LRTI-VAS) Scores [Mean (Standard Deviation); unit: score on a scale] — For each of the clinical symptoms of Lower Respiratory Tract Infections (LRTI; dyspnea, fatigue, cough, pain, and sputum), the participant assessed the severity using a 10 cm visual analogue scale (VAS) ranging from 0 = no symptoms to 10 = worst possible symptoms. A total LRTI score was calculated by summing up the score of each symptom (i.e., total LRTI score ranged from 0 to 50).
  score on a scale | 19.71 (9.74) | 14.87 (9.29) | 16.99 (9.65)
Baseline Quality of Life Questionnaire - Bronchiectasis (QOL-B) scale scores [Mean (Standard Deviation); unit: score on a scale] — The QOL-B questionnaire including 37 items on 8 scales (emotional functioning, health perceptions, physical functioning, respiratory symptoms, role functioning, social functioning, treatment burden, vitality) was used to assess particpant's quality of life (QoL). Each of the 37 items is scored from 1 to 4, and each of the 8 scale scores is standardised on a 0-100 point scale, with higher scores representing fewer symptoms or better functioning and QoL. Scales contain between 3 and 9 items, thus changing 1 answer category will correspond to a change of 11.1 to 3.7 points.
  score on a scale
    Emotional functioning | 83.97 (15.76) | 80.09 (13.14) | 81.72 (14.18)
    Health perceptions | 42.31 (24.41) | 52.31 (20.17) | 48.12 (22.23)
    Physical functioning | 58.46 (29.71) | 61.11 (28.21) | 60.00 (28.39)
    Respiratory symptoms | 60.01 (21.70) | 66.41 (12.75) | 63.72 (17.05)
    Role functioning | 62.05 (32.93) | 74.07 (23.97) | 69.03 (28.21)
    Social functioning | 59.83 (27.49) | 56.94 (26.97) | 58.15 (26.77)
    Treatment burden | 65.28 (17.25) | 73.61 (20.52) | 69.44 (18.81)
    Vitality | 41.03 (23.30) | 55.56 (19.80) | 49.46 (22.19)
Baseline Global Rating of Health (GRH) scores [Mean (Standard Deviation); unit: score on a scale] — Global Rating of Health was assessed as an interviewer questionnaire, which assesses global health as "excellent, good, fair or poor". For analysis, these were scored as 1 (poor) to 4 (excellent).
  score on a scale | 2.64 (0.84) | 2.78 (0.65) | 2.72 (0.73)
Body weight [Mean (Standard Deviation); unit: kilogram] | 52.24 (8.84) | 66.50 (14.40) | 60.26 (14.07)
Baseline 6-Minute Walking Distance (6MWD) [Mean (Standard Deviation); unit: meters] — The 6-minute walk test (6MWT) was performed in accordance with the European Respiratory Society/American Thoracic Society (ERS/ATS) guideline by technicians with documented training and experience. The 6MWT was performed twice at each visit.
  meters | 431.0 (89.6) | 440.8 (107.1) | 436.5 (98.4)
Baseline dyspnea scores [Mean (Standard Deviation); unit: score on a scale] — Participants scored the severity of dyspnea during a 6MWT using the Borg CR10 Scale. This was done before and immediately after each 6MWT. The post-walk score is reported below. Zero (0) on the scale corresponds to "nothing at all" and 10 to "extremely strong".
  score on a scale | 2.08 (2.48) | 2.47 (2.06) | 2.30 (2.22)
Baseline Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) [Mean (Standard Deviation); unit: percent predicted] — DLCO was assessed in accordance with the ERS/ATS task force standards using local, appropriately calibrated equipment. Parameters to be recorded are DLCO (absolute measured) and DLCO (predicted). The percent predicted DLCO is presented below. Two acceptable tests of DLCO were to be conducted and the average of these was used.
  percent predicted | 71.005 (23.076) | 73.166 (17.338) | 72.221 (19.926)
Baseline Forced Expiratory Volume in 1 Second (FEV1) [Mean (Standard Deviation); unit: percent predicted] — FEV1 was assessed in accordance with the ERS/ATS task force standards using local, appropriately calibrated equipment. Three valid measurements were made, and the highest value was used.
  percent predicted | 72.2231 (19.1010) | 69.7239 (24.2097) | 70.8173 (21.8175)
Baseline Forced Vital Capacity (FVC) [Mean (Standard Deviation); unit: percent predicted] — FVC was assessed in accordance with the ERS/ATS task force standards using local, appropriately calibrated equipment. Three valid measurements were made, and the highest value was used.
  percent predicted | 77.1785 (18.6934) | 82.7931 (22.0540) | 80.3367 (20.5249)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sputum Culture Conversion to Negative
Description: Sputum culture conversion is defined as at least 3 consecutive sputum samples without growth of NTM during the treatment period.
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Inhaled Molgramostim/Antimycobacterials: Inhaled molgramostim administered in participants who remain sputum culture positive while currently on a multidrug NTM-guideline based antimycobacterial regimen, which has been ongoing for at least 6 months prior to the Baseline Visit
  Inhaled molgramostim: 300 µg / dose molgramostim (recombinant human GM-CSF) for inhalation
  Antimycobacterial regimen: Multidrug NTM-guideline based antimycobacterial regimen
Arm/Group | Inhaled Molgramostim/Antimycobacterials | Inhaled Molgramostim
Number analyzed (Participants) | 14 | 18
Participants | 2 | 3

2. Secondary Outcome: Number of Participants With Sputum Smear Conversion to Negative
Description: Sputum smear conversion is defined as at least three consecutive negative acid-fast bacilli (AFB) stained sputum smears on microscopy during the treatment period among participants who were smear positive at Baseline.
Time Frame: 48 weeks
Population: Only participants who were smear positive at Baseline are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Molgramostim/Antimycobacterials | Inhaled Molgramostim
Number analyzed (Participants) | 13 | 16
Participants | 5 | 6

3. Secondary Outcome: Number of Participants With Durable Sputum Culture Conversion
Description: Durability is defined as sputum culture conversion at or before Week 24 and culture still negative for growth of NTM at 12-weeks follow-up.
Time Frame: 60 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Molgramostim/Antimycobacterials | Inhaled Molgramostim
Number analyzed (Participants) | 14 | 18
Participants | 1 | 1

4. Secondary Outcome: Number of Participants With Durable Sputum Smear Conversion
Description: Durability is defined as sputum smear conversion at or before Week 48 and AFB stained smear still negative for NTM at 12-weeks follow-up among participants who were smear positive at Baseline.
Time Frame: 60 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Molgramostim/Antimycobacterials | Inhaled Molgramostim
Number analyzed (Participants) | 14 | 18
Participants | 5 | 6

5. Secondary Outcome: Change From Baseline in Symptom Scores (Assessed Using Lower Respiratory Tract Infections - Visual Analogue Scale)
Description: For each of the clinical symptoms of Lower Respiratory Tract Infections (dyspnea, fatigue, cough, pain, and sputum), the participant assessed the severity using a 10 cm visual analogue scale (VAS) ranging from 0 = no symptoms to 10 = worst possible symptoms. A total LRTI score was calculated by summing up the score of each symptom (i.e., total LRTI score ranged from 0 to 50).
Time Frame: Baseline to Week 48
Population: Evaluable participants at Week 48 included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inhaled Molgramostim/Antimycobacterials | Inhaled Molgramostim
Number analyzed (Participants) | 9 | 16
score on a scale
  Total score | 2.48 (9.13) | 4.32 (13.32)
  Dyspnoea | 1.74 (2.50) | 0.91 (3.64)
  Tiredness | 1.29 (3.63) | 1.08 (3.96)
  Cough | 5.28 (3.08) | 3.35 (2.08)
  Color of phlegm | -1.88 (3.54) | 0.28 (2.24)
  Pain | 1.22 (2.76) | 0.58 (2.82)

6. Secondary Outcome: Change From Baseline in Symptom Scores (Assessed Using Quality of Life Questionnaire - Bronchiectasis (QOL-B))
Description: The QOL-B questionnaire including 37 items on 8 scales (emotional functioning, health perceptions, physical functioning, respiratory symptoms, role functioning, social functioning, treatment burden, vitality) was used to assess participant's quality of life (QoL). Each of the 37 items is scored from 1 to 4, and each of the 8 scale scores is standardised on a 0-100 point scale, with higher scores representing fewer symptoms or better functioning and QoL. Scales contain between 3 and 9 items, thus changing 1 answer category will correspond to a change of 11.1 to 3.7 points.
Time Frame: Baseline to Week 48
Population: Evaluable participants at Week 48 included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inhaled Molgramostim/Antimycobacterials | Inhaled Molgramostim
Number analyzed (Participants) | 9 | 16
score on a scale
  Emotional functioning | 0.00 (8.33) | 3.12 (12.12)
  Health perceptions | -12.96 (13.25) | -6.77 (21.99)
  Physical functioning | -17.78 (21.34) | -7.50 (28.38)
  Respiratory symptoms | -6.84 (8.24) | -4.34 (16.36)
  Role functioning | -13.33 (14.91) | -10.42 (22.96)
  Social functioning | -16.36 (15.43) | -7.81 (20.16)
  Treatment burden | -3.70 (12.83) | 4.44 (21.66)
  Vitality | -9.88 (12.96) | -7.64 (26.83)

7. Secondary Outcome: Change From Baseline in Global Rating of Health (GRH)
Description: GRH was assessed as an interviewer questionnaire, which assesses global health as "excellent, good, fair or poor". For analysis, these were scored as 1 (poor) to 4 (excellent).
Time Frame: Baseline to Week 48
Population: Evaluable participants at Week 48 included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inhaled Molgramostim/Antimycobacterials | Inhaled Molgramostim
Number analyzed (Participants) | 9 | 16
score on a scale | -0.78 (0.67) | -0.38 (0.81)

8. Secondary Outcome: Change From Baseline in Body Weight
Time Frame: Baseline to Week 48
Population: Evaluable participants at Week 48 included in the analysis.
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Inhaled Molgramostim/Antimycobacterials | Inhaled Molgramostim
Number analyzed (Participants) | 9 | 15
kilogram | -1.77 (2.51) | -1.44 (3.09)

9. Secondary Outcome: Change From Baseline in 6-Minute Walking Distance (6MWD)
Description: The 6-minute walk test (6MWT) was performed in accordance with the European Respiratory Society/American Thoracic Society (ERS/ATS) guideline by technicians with documented training and experience. The 6MWT was performed twice at each visit.
Time Frame: Baseline to Week 48
Population: Evaluable participants at Week 48 included in the analysis.
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Inhaled Molgramostim/Antimycobacterials | Inhaled Molgramostim
Number analyzed (Participants) | 9 | 15
meter | -17.1 (62.5) | 12.5 (56.2)

10. Secondary Outcome: Change From Baseline in Dyspnea Scores During a 6MWT
Time Frame: Baseline to Week 48
Population: Evaluable participants at Week 48 included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inhaled Molgramostim/Antimycobacterials | Inhaled Molgramostim
Number analyzed (Participants) | 9 | 15
score on a scale | 0.79 (0.92) | 1.43 (3.01)

11. Secondary Outcome: Number of Adverse Events (AEs) During the Trial Period
Description: All trial subjects were carefully monitored for the occurrence of AEs during the trial period from Baseline (Visit 2) to the 12-week Follow-up visit (Visit 15). AEs were collected by the investigator by a non-leading question and by reporting events directly observed or spontaneously volunteered by participants. Participants were also encouraged to contact the clinic in between visits if they experienced AEs or had any concerns.
Time Frame: 60 weeks
Measure: Number; unit: events
Arm/Group | Inhaled Molgramostim/Antimycobacterials | Inhaled Molgramostim
Number analyzed (Participants) | 14 | 18
events | 199 | 223

12. Secondary Outcome: Number of Serious AEs (SAEs) During the Trial Period
Description: SAEs were defined as any untoward medicinal occurrence or effect that at any dose:
  * Results in death
  * Is life-threatening
  * Requires hospitalisation or prolongation of existing hospitalisation
  * Results in persistent or significant disability or incapacity
  * Is a congenital abnormality or birth defect
  * May jeopardise the participant or may require medical intervention to prevent one or more of the outcomes listed above (Important Medical Events).
Time Frame: 60 weeks
Measure: Number; unit: events
Arm/Group | Inhaled Molgramostim/Antimycobacterials | Inhaled Molgramostim
Number analyzed (Participants) | 14 | 18
events | 14 | 17

13. Secondary Outcome: Number of Adverse Drug Reactions (ADRs) During the Trial Period
Description: All AEs were assessed by the investigator for causality (unlikely, possible, probable, not applicable) according to current regulatory standards. AEs which had a 'possible' or 'probable' causality were classified as ADRs.
Time Frame: 60 weeks
Measure: Number; unit: events
Arm/Group | Inhaled Molgramostim/Antimycobacterials | Inhaled Molgramostim
Number analyzed (Participants) | 14 | 18
events | 67 | 81

14. Secondary Outcome: Number of Severe AEs During the Trial Period
Description: All AEs were assessed by the investigator for severity (mild, moderate, severe) according to current regulatory standards.
Time Frame: 60 weeks
Measure: Number; unit: events
Arm/Group | Inhaled Molgramostim/Antimycobacterials | Inhaled Molgramostim
Number analyzed (Participants) | 14 | 18
events | 5 | 6

15. Secondary Outcome: Number of Participants Withdrawn From Treatment Due to an AE During the Trial Period
Time Frame: 60 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Molgramostim/Antimycobacterials | Inhaled Molgramostim
Number analyzed (Participants) | 14 | 18
Participants | 3 | 2

16. Secondary Outcome: Change From Baseline in Diffusing Capacity of the Lung for Carbon Monoxide (DLCO)
Time Frame: Baseline to Week 48
Population: Evaluable participants at Week 48 included in the analysis.
Measure: Mean (Standard Deviation); unit: percent predicted
Arm/Group | Inhaled Molgramostim/Antimycobacterials | Inhaled Molgramostim
Number analyzed (Participants) | 9 | 16
percent predicted | -4.565 (8.198) | -3.079 (7.766)

17. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) (% Predicted)
Time Frame: Baseline to Week 48
Population: Evaluable participants at Week 48 included in the analysis.
Measure: Mean (Standard Deviation); unit: percent predicted
Arm/Group | Inhaled Molgramostim/Antimycobacterials | Inhaled Molgramostim
Number analyzed (Participants) | 8 | 16
percent predicted | -1.7986 (10.2133) | -3.4011 (6.9830)

18. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) (% Predicted)
Time Frame: Baseline to Week 48
Population: Evaluable participants at Week 48 included in the analysis.
Measure: Mean (Standard Deviation); unit: percent predicted
Arm/Group | Inhaled Molgramostim/Antimycobacterials | Inhaled Molgramostim
Number analyzed (Participants) | 8 | 16
percent predicted | -2.4575 (6.6511) | -2.6135 (7.7040)

19. Secondary Outcome: Number of Subjects With Development of Anti-GM-CSF Antibodies in Serum
Description: Analyses for anti-GM-CSF antibodies were performed at a central laboratory.
Time Frame: 60 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Molgramostim/Antimycobacterials | Inhaled Molgramostim
Number analyzed (Participants) | 14 | 18
Participants | 5 | 10

ADVERSE EVENTS:
Time Frame: Baseline to 12-week follow-up (60 weeks in total).
Description: All trial subjects were carefully monitored for the occurrence of AEs during the trial period from Baseline (Visit 2) to the 12-week Follow-up visit (Visit 15). AEs were collected by the investigator by a non-leading question and by reporting events directly observed or spontaneously volunteered by participants. Participants were also encouraged to contact the clinic in between visits if they experienced AEs or had any concerns.
Arm/Group | Inhaled Molgramostim/Antimycobacterials | Inhaled Molgramostim
All-Cause Mortality (participants affected / at risk) | 2/14 | 1/18
Serious Adverse Events (participants affected / at risk) | 8/14 | 6/18
Other Adverse Events (participants affected / at risk) | 14/14 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Molgramostim/Antimycobacterials (N=14) | Inhaled Molgramostim (N=18)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Infective exacerbation of bronchiectasis (Infections and infestations) | 4 (5) | 3 (4)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1)
Lung infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Mycobacterium avium complex infection (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Molgramostim/Antimycobacterials (N=14) | Inhaled Molgramostim (N=18)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Fatigue (General disorders) | 4 (4) | 4 (7)
Pyrexia (General disorders) | 2 (4) | 4 (5)
Chest pain (General disorders) | 2 (2) | 2 (3)
Chest discomfort (General disorders) | 2 (2) | 2 (2)
Malaise (General disorders) | 1 (1) | 2 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Eosinophil count increased (Investigations) | 4 (4) | 6 (8)
C-reactive protein increased (Investigations) | 6 (6) | 3 (3)
Weight decreased (Investigations) | 1 (1) | 3 (3)
Blood creatinine increased (Investigations) | 1 (3) | 2 (2)
Blood urine present (Investigations) | 2 (3) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (15) | 13 (24)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 9 (10)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 (12) | 3 (8)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 4 (4)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 2 (3) | 4 (6)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (9) | 7 (13)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 5 (7)
Abdominal pain upper (Gastrointestinal disorders) | 2 (9) | 3 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Leukocyturia (Renal and urinary disorders) | 2 (3) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Infective exacerbation of bronchiectasis (Infections and infestations) | 4 (5) | 5 (9)
Upper respiratory tract infection (Infections and infestations) | 3 (5) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Mycobacterium avium complex infection (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
This was an exploratory study without hypothesis testing. Only descriptive statistics were used.

The study included participants with treatment refractory NTM infection, who were severely affected by their background disease (in most cases bronchiectasis). These participants probably had an even lower potential for improvement than was assumed prior to the study.

The study was further limited by the lack of a placebo control.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT03421743/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT03421743/SAP_001.pdf